CLINICAL TRIAL: NCT01960140
Title: Effects of Multiple Baricitinib (LY3009104) Doses on the Pharmacokinetics of a Cytochrome P450 3A Substrate, Simvastatin, in Healthy Subjects
Brief Title: A Study of Baricitinib and Simvastatin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14606; I4V-MC-JAGI (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — baricitinib; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin (Experimental): Single oral dose of 40 milligrams (mg) simvastatin on Day 1.
  Interventions: Drug: Simvastatin
- Baricitinib + Simvastatin (Experimental): Oral doses of 10 mg baricitinib once daily (QD) on Days 3 to 7, with a single oral dose of 40 mg simvastatin coadministered on Day 6.
  Interventions: Drug: Baricitinib; Drug: Simvastatin

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: Baricitinib + Simvastatin
Drug: Simvastatin — Administered orally

SUMMARY:
The purposes of this study are to determine the effects of baricitinib on the time it takes to remove simvastatin from the body and to look at how well-tolerated and safe baricitinib is when given alone and in combination with simvastatin. Side effects will be documented. The study will last approximately 7 days from the first dose to the end of the study (not including screening or follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Male participants - Agree to use 2 reliable methods of birth control with female partners of childbearing potential during the study and for at least 3 months following the last dose of study drug
* Female participants - Women not of childbearing potential due to surgical sterilization confirmed by medical history, or menopause
* Have a body mass index of 18.0 to 29.0 kilograms per meter squared (kg/m^2), inclusive
* Have clinical laboratory test results within the normal reference range
* Have normal renal function
* Have normal blood pressure and pulse rate

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving a study drug or off-label use of a drug or device, or are concurrently enrolled in any other type of medical research
* Have completed or discontinued within the last 90 days from a clinical trial involving a study drug
* Have previously completed or withdrawn from this study or any other study investigating baricitinib, and have previously received baricitinib
* Have known allergies to baricitinib, simvastatin, related compounds, or any components of the baricitinib or simvastatin formulations, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* Have a history of, or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (including hypothyroidism), hematological, or neurological disorders
* Have current or recent history of myalgia or muscle weakness
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Have a current or recent history of a clinically significant bacterial, fungal, parasitic, viral (not including rhinopharyngitis), or mycobacterial infection
* Have had symptomatic herpes zoster or herpes simplex infection within 90 days prior to the first dose
* Have an absolute neutrophil count (ANC) less than 2 × 10^9/liters (L) [2000 cells/microliter (μL)] at screening or day prior to first dose of study drug. For abnormal values, a single repeat will be allowed
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C infection and/or positive hepatitis C antibody
* Show evidence of hepatitis B infection and/or positive hepatitis B surface antigen
* Are women who are lactating
* Have been exposed to a live vaccine within 12 weeks prior to the first dose or expected to need/receive a live vaccine (including herpes zoster vaccination) during the course of the study
* Intend to use over-the-counter or prescription medication (including salicylate drugs) and/or herbal supplements within 14 days prior to dosing and during the study or intended use of vitamin supplements from Day 1 until discharge from the Clinical Research Unit (CRU)
* Have consumed or intend to consume grapefruit or grapefruit-containing products within 14 days prior to the first dose and throughout the study
* Have donated or lost blood of more than 500 milliliters (mL) within the last 3 months
* Have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females), or are unwilling to stop alcohol consumption from 48 hours prior to the first dose until discharge from the CRU at the end of Period 2
* History of, in the opinion of the investigator, excessive methylxanthine use within the previous 6 months, such as greater than (>)6 cups of coffee (or equivalent) per day
* Currently smoke more than 10 cigarettes per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leeds, West Yorkshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, fixed-sequence, 2-period study of healthy participants.
Groups:
- Simvastatin Then Baricitinib and Simvastatin: Period 1: 40-milligram (mg) tablet of simvastatin administered orally on Day 1.
  Period 2: 10-mg dose of baricitinib (2 × 4-mg and 1 × 2-mg tablets) administered orally once daily (QD) on Days 3 through 7, with coadministration of 40-mg simvastatin tablet on Day 6.
Period: Period 1 (Days 1-2)
Arm/Group | Simvastatin Then Baricitinib and Simvastatin
Started | 40
Received Simvastatin | 40
Completed | 40
Not Completed | 0
Period: Period 2 (Days 3-18)
Arm/Group | Simvastatin Then Baricitinib and Simvastatin
Started | 40
Received At Least 1 Dose of Baricitinib | 40
Received Simvastatin | 38
Completed | 38
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Simvastatin Then Baricitinib and Simvastatin: Period 1: 40-mg tablet of simvastatin administered orally on Day 1.
  Period 2: 10-mg dose of baricitinib (2 × 4-mg and 1 × 2-mg tablets) administered orally QD on Days 3 through 7, with coadministration of 40-mg simvastatin tablet on Day 6.
Arm/Group | Simvastatin Then Baricitinib and Simvastatin
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 40

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Simvastatin and Simvastatin Acid
Description: The Cmax of simvastatin [a cytochrome P450 (CYP) 3A substrate] and its active acid metabolite (simvastatin acid) is reported.
Time Frame: Period 1, Day 1 and Period 2, Day 6: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 and 48 hours postdose
Population: Participants who received study drug (simvastatin in Period 1 and at least 1 dose of baricitinib and simvastatin in Period 2) and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Simvastatin: Period 1: 40-mg tablet of simvastatin administered orally on Day 1.
- Baricitinib and Simvastatin: Period 2: 10-mg dose of baricitinib (2 × 4-mg and 1 × 2-mg tablets) administered orally QD on Days 3 through 7, with coadministration of 40-mg simvastatin tablet on Day 6.
Arm/Group | Simvastatin | Baricitinib and Simvastatin
Number analyzed (Participants) | 40 | 38
nanograms per milliliter (ng/mL)
  Simvastatin | 6.85 (74) | 4.65 (57)
  Simvastatin Acid | 1.93 (68) | 1.60 (50)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Zero to Infinity [AUC(0-∞)] of Simvastatin and Simvastatin Acid
Description: The AUC(0-∞) of simvastatin (a CYP3A substrate) and its active acid metabolite (simvastatin acid) is reported.
Time Frame: Period 1, Day 1 and Period 2, Day 6: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24 and 48 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | Simvastatin | Baricitinib and Simvastatin
Number analyzed (Participants) | 39 | 36
nanograms*hour/milliliter (ng*h/mL)
  Simvastatin (n=39, 36) | 40.7 (86) | 33.7 (75)
  Simvastatin Acid (n=33, 32) | 26.4 (81) | 21.0 (64)

ADVERSE EVENTS:
Time Frame: Baseline through study completion (up to Day 18)
Groups:
- Simvastatin: A 40-mg tablet of simvastatin administered orally on Day 1.
  Adverse events (AEs) are reported from baseline through predose on Day 3.
- Baricitinib: A 10-mg dose of baricitinib (2 × 4-mg and 1 × 2-mg tablets) administered orally QD on Days 3 through 5.
  AEs are reported postdose on Day 3 through predose on Day 6.
- Baricitinib and Simvastatin: A 10-mg dose of baricitinib (2 × 4-mg and 1 × 2-mg tablets) administered orally QD on Days 6 and 7, with coadministration of 40-mg simvastatin tablet on Day 6.
  AEs are reported postdose on Day 6 up to Day 18.
Arm/Group | Simvastatin | Baricitinib | Baricitinib and Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 3/40 | 1/40 | 3/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=40) | Baricitinib (N=40) | Baricitinib and Simvastatin (N=38)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (4) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days